CLINICAL TRIAL: NCT03682588
Title: A Functional Exercise Program Improves Pain and Health Related Quality of Life in Patients With Fibromyalgia: A Randomized Controlled Trial
Brief Title: A Functional Exercise Program Improves Pain and Health Related Quality of Life in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Giovana Fernandes, PhD Student, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 719.779
Record Dates: First submitted 2018-08-03; First posted 2018-09-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Exercise; Functional training
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Randomised electronically generated randomisation table. Secret allocation (sealed opaque envelopes).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional exercise group (Experimental): Functional exercise program with 14 exercises, two times/week, during 14 weeks. Two sets of 10 repetitions each, with 30 seconds interval.
  Interventions: Other: Physical activity
- Stretching exercise group (Active Comparator): Stretching exercise program with 17 exercises, two times/week, during 14 weeks and each movement was repeated by three times and held for 20 seconds each
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Physical activity — The Functional exercise group performed functional exercise training for 45 minutes twice a week for 14 weeks. The Stretching exercise group performed stretching exercises with the same duration and frequency.
  Other Names: Functional exercise group and Stretching exercise group

SUMMARY:
Fibromyalgia is a syndrome characterized mainly by chronic generalized pain that affects the physical fitness and functional capacity of patients. There is increasing evidence of the benefits of physical exercise in improving fibromyalgia symptoms, making these interventions part of therapeutic arsenal. Objective: To evaluate the effectiveness of a program of functional exercises in reducing pain, improving functional capacity, increasing muscle strength, improving flexibility, balance and quality of life of patients with fibromyalgia. Intervention: The intervention group performed functional physical training for 45 minutes twice a week for 14 weeks. The control group will perform stretching exercises with the same duration and frequency. evaluation instruments: Visual Analog Scale for pain; Fibromyalgia Impact Questionnaire; Time-up and go test; 1Repetitian Maximum test; Sit and reach test; Berg Balance Scale; and Short Form-36 and amount of analgesics used during the intervention period was evaluated.

DETAILED DESCRIPTION:
Fibromyalgia is a syndrome characterized mainly by chronic generalized pain that affects the physical fitness and the functional capacity of patients. There is growing evidence of the benefits of exercise to improve fibromyalgia symptoms, making these interventions part of the therapeutic arsenal. Objective: To evaluate the effectiveness of a functional exercise program in reducing pain, improving functional capacity, increasing muscle strength, improving flexibility, balance and quality of life of patients with fibromyalgia. METHODS: This was a randomized controlled trial with blind evaluator. 82 female patients with fibromyalgia were included, aged between 18 and 65 years, randomized into two groups, intervention and control. The intervention group performed functional physical training for 45 minutes twice a week for 14 weeks. The control group performed stretching exercises with the same duration and frequency. The evaluation instruments were: Visual Analog Scale for pain evaluation; Fibromyalgia Impact Questionnaire, to evaluate health-related quality of life; Time-up and go test for functional performance assessment; 1Repetitium Maximum, for evaluation of muscle strength; sit and reach test for the assessment of flexibility; Berg Balance Scale, to assess balance; and Short Form-36 to assess overall quality of life. In addition, the amount of analgesics used during the intervention period was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Classification of fibromyalgia based on the criteria of the American College of Rheumatology
* Age 18 to 65 years;
* Pain intensity between 4 and 8cm on a visual analog scale ranging from 0 to 10cm
* Stable medication for at least three months

Exclusion Criteria:

* Uncontrolled cardiorespiratory disease
* Health condition for which physical exercise was contraindicated
* Serious psychiatric disorder
* Uncontrolled diabetes mellitus
* Inflammatory rheumatic disease
* History of regular physical exercise (30min, 3 times a week) in the previous 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2020-01-06 (Actual)

PRIMARY OUTCOMES:
Change in pain | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the Visual Analogue Scale for pain. Scores ranges from 0 to 10 with higher values represent a worse pain.

SECONDARY OUTCOMES:
Change in Muscular Strength | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the one-repetition maximum test
Change in functional performance | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the Time-up and go test
Change in balance | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the Berg balance scale to evaluate balance. Scores ranges from 0 to 56 with higher values represent a worse balance.
Change in Flexibility | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the sit and reach test (Wells Bench)
Change in General quality of life | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the Short-form 36 questionnaire for quality of life. Scores ranges from 0 to 100 with higher values represent a better quality of life..
Change in medications consumption | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated the amount of acetominophen (500mg de 6/6 hours) used for pain
Change in health-related quality of life | Baseline, after 7, 14, 26 and 38 weeks
  Evaluated using the Fibromyalgia Impact Questionnaire. Scores ranges from 0 to 100 with higher values represent a worse quality of life..

CONTACTS AND LOCATIONS:
Overall Officials: Jamil Natour, Professor, Study Director — Federal University of São Paulo
Locations (1):
- Rheumatology outpatient clinics of a university hospital;, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Fernandes G, Nery M, Meireles SM, Santos R, Natour J, Jennings F. A functional exercise program improves pain and health related quality of life in patients with fibromyalgia: a randomized controlled trial. Adv Rheumatol. 2024 Oct 24;64(1):81. doi: 10.1186/s42358-024-00422-7. PMID 39449056